CLINICAL TRIAL: NCT02611115
Title: Optimizing Tube Voltage Settings and Injection Parameters for the Individual Patient in CT Pulmonary Angiography.
Brief Title: Optimizing Protocols for the Individual Patient in CT Pulmonary Angiography.
Acronym: OptIPeCT
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Marco Das, MD, PhD, Maastricht University Medical Center
Other Study IDs: 15-4-167
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Multidetector Computed Tomography; Radiation Dosage; Contrast Media; Individualized Medicine
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Computed tomographic pulmonary angiography (CTPA) is considered the gold standard for the diagnosis of pulmonary embolism (PE). PE is a potentially fatal disease in which a thrombus is lodged into a pulmonary artery blocking blood flow and potentially leading to respiratory distress, acute right cardiac failure or death. Therefore early and correct diagnosis is crucial.

The diagnostic and clinical value of CTPA has already been firmly substantiated. Unfortunately up to 7.3% of PE scans are still deemed to be non-diagnostic, for example due to insufficient contrast enhancement in the target arteries.

Therefore future research should focus on two important aspects of CT imaging. On the one hand optimal enhancement for the individual patient, on the other hand preventing additional risk of CT imaging - namely contrast induced nephropathy (CIN) and radiation risk. Thus the purpose of our study will be to optimize radiation dose settings (e.g. tube voltage, tube current) and CM application for the individual patient in CTPA.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of pulmonary embolism

Exclusion Criteria:

* Severe allergy against Iopromide or any of the ingredients, previous severe CM reaction (according to current ESUR guidelines), renal insufficiency, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for CTPA with a clinical suspicion of pulmonary embolism will be included.
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Image quality | one year
  Evaluation of subjective and objective image quality based on individualized CTPA protocols

SECONDARY OUTCOMES:
Reduction of radiation dose | one year
  Effect of individualized tube voltage settings on radiation

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands